CLINICAL TRIAL: NCT04887857
Title: A Phase 1B, Open-label, Global, Multicenter, Dose Determination Study to Evaluate Safety, Tolerability, and Preliminary Efficacy of CC-486 (ONUREG®) in Combination Therapy in Subjects With Acute Myeloid Leukemia (AML)
Brief Title: A Study to Assess Safety and Tolerability of CC-486 (ONUREG®, Oral Azacitidine) in Combination Therapy in Participants With Acute Myeloid Leukemia (AML)
Acronym: OMNIVERSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-486-AML-004; 2020-004941-35 (EudraCT Number)
Expanded Access: NCT03723135 (Approved for marketing)
Record Dates: First submitted 2021-05-11; First posted 2021-05-14 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Acute Myeloid Leukemia; CC-486; Onureg; oral azacitidine; venetoclax; Venclexta; Venclyxto
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — cc-486; Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CC-486 in combination with Venetoclax (Experimental)
  Interventions: Drug: CC-486; Drug: Venetoclax

INTERVENTIONS:
Drug: CC-486 — Specified dose on specified days
  Other Names: ONUREG®, oral azacitidine
Drug: Venetoclax — Specified dose on specified days
  Other Names: VENCLEXTA®, VENCLYXTO®

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and preliminary efficacy of CC-486 (ONUREG®) in combination with venetoclax in relapsed and/or refractory Acute Myeloid Leukemia (AML) and newly diagnosed AML.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of the following for Acute Myeloid Leukemia (AML)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2. ECOG 3 is allowed if participants are 18 to 74 years old with comorbidities
* Agree to serial bone marrow aspirate/biopsies

Exclusion Criteria:

* Suspected or proven to have acute promyelocytic leukemia based on morphology, immunophenotype, molecular assay, or karyotype
* Received prior hypomethylating agent (HMA) therapy for myelodysplastic syndromes/Chronic myelomonocytic leukemia then develop AML within 4 months of discontinuing the HMA therapy
* Prior history of malignancy unless the participant has been free of the disease for ≥ 1 year prior to the start of study treatment

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 42 days after first dose
Incidence of type of adverse events (AEs) | From informed consent form (ICF) signature to 28 days after last dose of study drug
Incidence of frequency of AEs | From informed consent form (ICF) signature to 28 days after last dose of study drug
Incidence of severity of AEs | From informed consent form (ICF) signature to 28 days after last dose of study drug
Incidence of relationship of AEs to study treatment | From informed consent form (ICF) signature to 28 days after last dose of study drug
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | From informed consent form (ICF) signature to 28 days after last dose of study drug
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | From informed consent form (ICF) signature to 28 days after last dose of study drug
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | From informed consent form (ICF) signature to 28 days after last dose of study drug

SECONDARY OUTCOMES:
Rate of complete remission (CR)/complete remission with partial hematologic recovery (CRh) | Up to approximately 12 months
Overall Response Rate (ORR) | Up to approximately 12 months
Minimal Residual Disease (MRD) Response Rate | Up to approximately 12 months
MRD Conversion Rate | Up to approximately 12 months
Rate of complete remission (CR)/complete remission with incomplete recovery of blood counts (CRi) | Up to approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- United States (8):
  - Local Institution - 104, Stanford, California
  - Local Institution - 110, Denver, Colorado
  - Local Institution - 105, Boston, Massachusetts
  - Local Institution - 106, New York, New York
  - Local Institution - 113, New York, New York
  - Local Institution - 102, Cleveland, Ohio
  - Local Institution - 111, Oklahoma City, Oklahoma
  - Local Institution - 101, Houston, Texas
- Australia (2):
  - Local Institution - 202, North Melbourne, Victoria
  - Local Institution - 201, Melbourne

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT04887857.html